CLINICAL TRIAL: NCT01124279
Title: A Phase I, Randomized, Open-Label, Single-Dose, 2-Part, 4-Treatment, 4-Way Crossover Study in Healthy Adult Subjects to Evaluate the Pharmacokinetics of Various AMG 853 Formulations When Administered Under Fasted and Fed Conditions
Brief Title: Single-dose, Pharmacokinetics of AMG 853 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20090226
Record Dates: First submitted 2010-05-13; First posted 2010-05-17 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Healthy Volunteers
Keywords: Amgen; Healthy; Adult
MeSH Terms: interventions — vidupiprant

ARMS (1):
- AMG 853 (Experimental)
  Interventions: Drug: AMG 853

INTERVENTIONS:
Drug: AMG 853 — Single dose administration of AMG 853 in tablet form to healthy adult subjects

SUMMARY:
To determine the bioavailability and the effect of food on the pharmacokinetics under fasted and fed conditions

ELIGIBILITY:
Inclusion Criteria:

* Non-nicotine or tobacco using, healthy male and/or female subjects between 18 and 55 years of age, inclusive, with no history or evidence of clinically relevant medical disorders as determined by the investigator in consultation with the Amgen physician
* Females must be of non-reproductive potential (ie, postmenopausal by history - no menses for 1 year - and FSH consistent with postmenopausal status per laboratory ranges; or history of hysterectomy; or history of bilateral tubal ligation; or history of bilateral oophorectomy).
* Physical examination, clinical laboratory test values and ECGs are clinically acceptable to the investigator and Amgen.
* Males must agree to use highly effective methods of birth control for the duration of the study and continuing for 12 weeks after the last dose of AMG 853. Highly effective methods of birth control (i.e., those with a failure rate of less than 1% per year) include sexual abstinence, vasectomy or a condom supplemented with the use of a spermicide, where available, in combination with one of the following methods used by the female partner: in regions where spermicide is available, diaphragm or cervical/vault caps supplemented with spermicide, hormonal birth control (implants, injectables, or combined oral contraceptives), intrauterine devices (IUDs).
* Male subjects whose partners become pregnant during the study will not receive subsequent scheduled doses, must practice sexual abstinence or use a condom for two weeks following the last dose, and will be followed for safety through end of study. The pregnant partner information will be reported to Amgen as per the Pregnancy Notification Worksheet.
* Body mass index between 18 and 30 kg/m2, inclusive.

Exclusion Criteria:

* History or evidence of clinically significant disorder, condition or disease that, in the opinion of the investigator or Amgen physician, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion.
* Creatinine clearance within the screening period of less than 80 mL/min as calculated by the Cockcroft-Gault method.
* History suggestive of esophageal, gastric, or duodenal ulceration or bowel disease (including but not limited to peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease, or irritable bowel syndrome), or a history of gastrointestinal surgery other than uncomplicated appendectomy.
* Any positive test for cotinine (tobacco use) on the day before dosing of each treatment period (day -1, 7, 14 and 21). A positive cotinine level is defined as any level exceeding the upper limit of normal per local laboratory reference ranges.
* Known substance abuse (eg, alcohol, licit or illicit drugs) within 1 year of dosing.
* Any positive test for drugs and or alcohol use on the day before dosing of each treatment period (day -1, 7, 14 and 21). Alcohol should not be consumed within 48 hours of day -1 and throughout the study.
* Females who are lactating/breastfeeding.
* Males with pregnant partners.
* Subjects who require specialized diets or have dietary restrictions that would prevent them from complying with the study requirements.
* Inability or unwillingness to swallow tablets.
* Unwilling to consume a standardized high-fat breakfast (approximately 800 to 1000 calories) consisting of approximately 33 g protein, 58 g carbohydrate, and 75 g fat, respectively (e.g. 2 eggs fried in butter, 2 strips of bacon, 2 slices of toast with butter, 4 ounces of hash-brown potatoes, and 8 ounces of whole milk).
* Subjects who are lactose intolerant
* A history of malignancy of any type, other than surgically excised non-melanomatous skin cancers or in situ cervical cancer within 5 years before the day of dosing.
* Donated greater than 500 mL of blood or blood products within 60 days of dosing.
* Receiving or has received any investigational drug (or using or has used an investigational device) within the 30 days before receiving the first dose of study medication, or at least 5 elimination half-lives (whichever is longer).
* Subjects who were previously exposed to AMG 853.
* Use of any over-the-counter or prescription medications (specifically including, but not limited to, antacids, H2- blockers, and proton pump inhibitors, aspirin or other non-steroidal anti-inflammatory drugs [NSAIDS]) within 30days of dosing. Acetaminophen (up to 2 g per day) for analgesia and hormone replacement therapy (eg, estrogen) will be allowed.
* Use of any known inhibitors of CYP3A4/P-gp such as ketoconazole, itraconazole, HIV protease inhibitors, nefazadone, cyclosporine, erythromycin, clindamycin, tetracycline, and clarithromycin within 14 days or 5 half lives, which ever is longer; or grapefruit juice or grapefruit containing products within 7 days prior to investigational product administration.
* Use of any known CYP inducers such as rifampin, corticosteroids, or anticonvulsants within 30 days or 5 half-lives, which ever is longer, before investigational product administration.
* Use of any herbal medicine (eg, St. John's wort) within 30 days before investigational product administration. All herbal medicines, vitamins, and supplements consumed by the subject within 30 days prior to the first dose of investigational product and continued use, if appropriate, will be reviewed by the Principal Investigator and the Amgen Medical Monitor.
* History of hypersensitivity or allergic reaction to sulfonamide drugs.
* Positive for HIV antibodies, hepatitis B surface antigen, or hepatitis C antibodies.
* Known history of Gilbert's syndrome.
* Any other condition that might reduce the chance of obtaining data (eg, known poor compliance) required by the protocol or that might compromise the ability to give truly informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | throughout study duration

SECONDARY OUTCOMES:
Treatment-emergent adverse events, safety and laboratory assessments | throughout study duration

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com